CLINICAL TRIAL: NCT03783078
Title: A Phase 3 Open-label, Single Arm Study to Evaluate the Safety and Efficacy of Pembrolizumab (MK-3475) as First Line Therapy in Participants With Advanced Merkel Cell Carcinoma (KEYNOTE-913)
Brief Title: Pembrolizumab (MK-3475) as First-line Therapy for Advanced Merkel Cell Carcinoma (MK-3475-913)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-913; MK-3475-913 (Other: MSD); KEYNOTE-913 (Other: MSD); 2018-002601-57 (EudraCT Number)
Record Dates: First submitted 2018-12-19; First posted 2018-12-20 (Actual); Results first posted 2023-02-17 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Merkel Cell Carcinoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2); Merkel cell carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab (MK-3475) 200 mg (adult participants) or 2 mg/kg (up to 200 mg; pediatric participants) on Day 1 of each 3-week cycle (Q3W) intravenous (IV), for up to 35 administrations (approximately 2 years)
  Interventions: Drug: Pembrolizumab (MK-3475)

INTERVENTIONS:
Drug: Pembrolizumab (MK-3475) — 200 mg (adult participants) or 2 mg/kg (up to 200 mg; pediatric participants) on Day 1 of each 3-week cycle (Q3W) IV up to 35 administrations (approximately 2 years).
  Other Names: MK-3475

SUMMARY:
This is a single-arm, open-label, multicenter, efficacy, and safety study of pembrolizumab in adult and pediatric participants with previously untreated advanced Merkel Cell Carcinoma (MCC). The primary objective of the trial is to assess the objective response rate, as assessed by blinded independent central review per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, following administration of pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female and at least 12 years of age, at the time of signing the informed consent/assent.
* Have histologically confirmed diagnosis of locoregional MCC that has recurred following standard locoregional therapy with surgery and/or radiation therapy and is not amenable to local therapy or metastatic MCC (Stage IV) as per American Joint Committee on Cancer (AJCC) 8th edition guidelines.
* Have been untreated for advanced or metastatic disease except as follows:

  1. Prior intratumoral therapy will be permitted.
  2. Prior adjuvant or neoadjuvant therapy containing systemic chemotherapy will be permitted if treatment concluded at least 3 months prior to Cycle 1 Day 1 (C1D1).
  3. Prior adjuvant or neoadjuvant therapy containing anti-PD-1/L1 or anti-CTLA-4 (cytotoxic T-lymphocyte-associated protein 4) therapy will not be permitted.
* Have at least 1 measurable lesion by computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST 1.1 criteria as determined by the local site investigator/radiology assessment.
* Toxic effect(s) of the most recent prior therapy have resolved to Grade 1 or less (except alopecia).
* Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:
* Is not a woman of childbearing potential (WOCBP)
* OR
* Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis).
* A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 72 hours before the first dose of study intervention.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 or Lansky Play-Performance Scale (LPS) ≥50 for pediatric participants up to and including 16 years of age.
* Have adequate organ function

Exclusion Criteria:

* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years with certain exceptions.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis with certain exceptions.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to C1D1.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease-modifying agents, corticosteroids or immunosuppressive drugs).
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
* Has a known history of active tuberculosis (TB; Bacillus tuberculosis).
* Has clinically significant cardiac disease within 6 months of C1D1, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
* Has not received standard locoregional therapy with surgery and/or radiation therapy for the treatment of local or locoregional disease. Note: This exclusion criterion does not apply to participants who are diagnosed with unresectable or metastatic MCC.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor.
* Has received prior systemic anticancer therapy including investigational agents within 12 weeks prior to C1D1.
* Has received radiotherapy within 2 weeks prior to start of study intervention.
* Has received a live vaccine within 30 days prior to C1D1.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to C1D1.
* Has had an allogenic tissue/solid organ transplant.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2024-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (22):
- United States (2):
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone Health ( Site 0006), New York, New York
  - Icahn School of Medicine at Mount Sinai ( Site 0004), New York, New York
- Australia (2):
  - Melanoma Institute Australia ( Site 0400), North Sydney, New South Wales
  - Calvary Mater Newcastle ( Site 0402), Waratah, New South Wales
- Canada (2):
  - Moncton Hospital - Horizon Health Network ( Site 0055), Moncton, New Brunswick
  - Princess Margaret Cancer Centre ( Site 0051), Toronto, Ontario
- France (5):
  - Hopital de la Cote de Nacre - Caen ( Site 0204), Caen, Calvados
  - CHU de Bordeaux- Hopital Saint Andre ( Site 0203), Bordeaux, Gironde
  - Hopital Ambroise Pare Boulogne ( Site 0201), Boulogne-Billancourt, Hauts-de-Seine
  - C.H.R.U. de Tours. Hopital Trousseau ( Site 0202), Chambray-lès-Tours, Indre-et-Loire
  - CHRU Lille - Hopital Claude Huriez ( Site 0200), Lille, Nord
- Italy (4):
  - Azienda Ospedaliera Universitaria Senese ( Site 0224), Siena, Tuscany
  - IEO Istituto Europeo di Oncologia ( Site 0223), Milan
  - Istituto Nazionale Tumori Fondazione Pascale ( Site 0222), Napoli
  - Istituto Oncologico Veneto ( Site 0221), Padua
- Auckland City Hospital ( Site 0427), Auckland, New Zealand
- Spain (4):
  - Hospital General Universitario de Valencia ( Site 0262), Valencia, Valenciana, Comunitat
  - Hospital Universitari Vall d Hebron ( Site 0264), Barcelona
  - Hospital Clinic de Barcelona ( Site 0261), Barcelona
  - Hospital Universitario La Paz ( Site 0263), Madrid
- Sweden (2):
  - Karolinska Universitetssjukhuset Solna ( Site 0281), Solna, Stockholm County
  - Sahlgrenska Universitetssjukhuset ( Site 0282), Gothenburg, Västra Götaland County

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Mortier L, Villabona L, Lawrence B, Arance A, Butler MO, Beylot-Barry M, Saiag P, Samimi M, Ascierto PA, Spada F, De Pontville M, Maio M, Berrocal A, Espinosa E, Capdevila J, Levin M, Das D, Krepler C, Grebennik D, Chiarion-Sileni V. Pembrolizumab for the First-Line Treatment of Recurrent Locally Advanced or Metastatic Merkel Cell Carcinoma: Results from the Single-Arm, Open-Label, Phase III KEYNOTE-913 Study. Am J Clin Dermatol. 2024 Nov;25(6):987-996. doi: 10.1007/s40257-024-00885-w. Epub 2024 Oct 8. PMID 39377880
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26661&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants of at least 12 years of age with advanced Merkel cell carcinoma (MCC) were recruited to evaluate the safety and efficacy of Pembrolizumab (MK-3475) as first-line therapy.
Groups:
- Pembrolizumab 200 mg: Adult participants received pembrolizumab (MK-3475) 200 mg or pediatric participants received 2 mg/kg (up to 200 mg) on Day 1 of each 3-week cycle (Q3W) intravenously (IV), for up to 35 administrations (approximately 2 years).
Period: Overall Study
Arm/Group | Pembrolizumab 200 mg
Started | 55
Completed | 0
Not Completed | 55
Not completed — Death | 31
Not completed — Sponsor Decision | 23
Not completed — Withdrawal by Parent/Guardian | 1

BASELINE CHARACTERISTICS:
Groups:
- Pembrolizumab 200 mg: Adult participants received pembrolizumab (MK-3475) 200 mg or pediatric participants received 2 mg/kg (up to 200 mg) on Day 1 Q3W IV for up to 35 administrations (approximately 2 years).
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 39
  More than one race | 0
  Unknown or Not Reported | 16

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). The percentage of participants who experienced CR or PR as assessed by blinded independent central review (BICR) were presented.
Time Frame: Up to ~34 months
Population: The analysis population consisted of all allocated participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 55
Percentage of participants | 49.1 [35.4 to 62.9]

2. Secondary Outcome: Duration of Response (DOR)
Description: For participants who demonstrated a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR was defined as the time from first documented evidence of a CR or PR until progressive disease (PD) or death. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions as well as an absolute increase of at least a 5 mm in the sum of diameters. The appearance of one or more new lesions was also considered PD. DOR assessments were based on BICR with confirmation. The DOR as assessed using RECIST 1.1 for all participants who experienced a confirmed CR or PR was presented.
Time Frame: Up to ~58 months
Population: The analysis population consisted of all allocated participants who received at least 1 dose of study treatment, and who experienced a confirmed CR or confirmed PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 27
Months | 39.8 [23.8 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse.

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-Free Survival was defined as the time from the first dose of study treatment to the first documented evidence of disease progression per RECIST 1.1 by BICR or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. PFS as assessed by BICR per RECIST 1.1 was presented.
Time Frame: Up to ~58 months
Population: The analysis population consisted of all allocated participants who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 55
Months | 9.3 [3.0 to 25.5]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the first dose of study treatment until death from any cause.
Time Frame: Up to ~58 months
Population: The analysis population consisted of all allocated participants who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 55
Months | 24.3 [12.4 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event

5. Secondary Outcome: Number of Participants With One or More Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants with at least one AE was assessed.
Time Frame: Up to ~58 months
Population: The analysis population consisted of all allocated participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 55
Participants | 52

6. Secondary Outcome: Number of Participants Who Discontinued From Study Treatment Due to an AE
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued from study treatment due to an AE was assessed.
Time Frame: Up to ~27 months
Population: The analysis population consisted of all allocated participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 55
Participants | 18

ADVERSE EVENTS:
Time Frame: Up to ~58 months
Description: All-cause mortality includes all allocated participants. AEs include participants who received ≥1 dose of study treatment. Per protocol, disease progression was not considered an AE, unless related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study treatment were excluded as AEs.
Arm/Group | Pembrolizumab 200 mg
All-Cause Mortality (participants affected / at risk) | 32/55
Serious Adverse Events (participants affected / at risk) | 24/55
Other Adverse Events (participants affected / at risk) | 49/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 200 mg (N=55)
Colitis (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Empyema (Infections and infestations) | 1 (1)
Encephalitis (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (11)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (9)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 200 mg (N=55)
Anaemia (Blood and lymphatic system disorders) | 9 (11)
Vertigo (Ear and labyrinth disorders) | 3 (4)
Hyperthyroidism (Endocrine disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Constipation (Gastrointestinal disorders) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 7 (11)
Dry mouth (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 8 (10)
Vomiting (Gastrointestinal disorders) | 5 (5)
Asthenia (General disorders) | 11 (20)
Fatigue (General disorders) | 14 (18)
Oedema peripheral (General disorders) | 5 (5)
Pyrexia (General disorders) | 7 (9)
COVID-19 (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 3 (6)
Fall (Injury, poisoning and procedural complications) | 3 (4)
Alanine aminotransferase increased (Investigations) | 10 (13)
Amylase increased (Investigations) | 5 (6)
Aspartate aminotransferase increased (Investigations) | 12 (14)
Blood alkaline phosphatase increased (Investigations) | 4 (4)
Blood creatine phosphokinase increased (Investigations) | 3 (4)
Blood creatinine increased (Investigations) | 4 (4)
Lipase increased (Investigations) | 10 (11)
Weight decreased (Investigations) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 6 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (11)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5)
Dysgeusia (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 6 (7)
Insomnia (Psychiatric disorders) | 3 (3)
Dysuria (Renal and urinary disorders) | 3 (3)
Haematuria (Renal and urinary disorders) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Eczema (Skin and subcutaneous tissue disorders) | 5 (6)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (19)
Rash (Skin and subcutaneous tissue disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT03783078/Prot_SAP_000.pdf